CLINICAL TRIAL: NCT04616274
Title: Pharmacokinetics of Venetoclax in Patients With Chronic Lymphocytic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006213RINC
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Venetoclax: Adult CLL patients (≥ 20 year-old) who have already initiated or are going to receive venetoclax treatment at National Taiwan University Hospital/National Taiwan University Cancer Center from July 2020 to December 2025.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — This prospective study will draw blood from every patient to measure the venetoclax blood concentration. After blood concentration analysis by ultra-high performance liquid chromatography tandem mass spectrometry (UHPLC-MS/MS), the investigator will report the concentration to clinicians.

SUMMARY:
Venetoclax is a treatment for chronic lymphocytic leukemia (CLL) and acute myeloid leukemia (AML). However, the pharmacokinetic data in Chinese population, as well as the change of venetoclax plasma concentration while taking CYP enzyme inducers or inhibitors, remained unknown so far. Therefore, the aim of this study is to investigate the pharmacokinetic characteristics of venetoclax.

DETAILED DESCRIPTION:
Venetoclax has been approved for treatment of adult patients with chronic lymphocytic leukemia (CLL). Currently, there is not enough data of CLL populations from Chinese or other Asian regarding its efficacy or adverse reactions. In the phase 3 MURANO trial (NCT02005471), only 8 Asians (2.06%) were included, while other phase 1 or phase 2 studies did not show the percentage of Asian population. According to a venetoclax population pharmacokinetic study published in 2016, which integrated 505 subjects from 8 clinical trials, concluded that race was not a covariate that affect venetoclax PK. However, only 6 Asians (1.19%) were included, and some of the subjects were small lymphocytic lymphoma (SLL), non-Hodgkin's lymphoma (NHL) or healthy volunteers.

The pharmacokinetics of venetoclax is affected by many factors, and the most influential factors may be fat content from dietary and concomitant use of CYP3A inhibitors or inducers. In particular, patients with hematological malignancies often require antifungal agents (such as voriconazole, posaconazole) as prophylaxis or treatment of fungal infections during chemotherapy. Therefore, these two factors will be considered in this study.

The most common side effect after using venetoclax is neutropenia. About 60.8% of patients developed any grades neutropenia, 43.3% required dose interruption, 8.2% required dosage reduction, and 2.6% required permanent treatment discontinuation because of neutropenia in phase 3 MURANO trial. Recent studies have found that the probability of ≥ grade 3 neutropenia and infection seems to be inversely related to the blood concentration of venetoclax, that is, the higher the blood concentration of venetoclax, the lower the probability of neutropenia and infection.

This observational study is designed to examine the plasma concentration of venetoclax in patients with CLL or AML, to create a pharmacokinetic model of venetoclax in Chinese population, and to analyze the extent to which CYP enzyme inhibitors and inducers may have effect on venetoclax plasma concentration. Moreover, the association between therapeutic effectiveness, adverse events, and venetoclax plasma concentration will also be analyzed in this study, and the final purpose is to establish the principle of clinical dose adjustment in the future.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 20 year-old) with diagnosis of chronic lymphocytic leukemia
* Patients who meet the above criteria and have already initiated or are going to receive venetoclax treatment at National Taiwan University Hospital/National Taiwan University Cancer Center from July 2020 to December 2025

Exclusion Criteria:

* Patients who are unable to cooperate with blood drawing
* Patients who have not submit the informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult chronic lymphocytic leukemia patients (≥ 20 year-old) who have already initiated or are going to receive venetoclax treatment at National Taiwan University Hospital/National Taiwan University Cancer Center from August 2020 to December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under curve (AUC) of venetoclax in Chinese population | July 1, 2020 to December 31, 2025
  Area under curve (AUC) will be calculated through multiple plasma concentrations drawn from the patients after taking venetoclax.
Half-life (T1/2) of venetoclax in Chinese population | July 1, 2020 to December 31, 2025
  Half-life (T1/2) will be calculated through multiple plasma concentrations drawn from the patients after taking venetoclax.
Clearance (CL) of venetoclax in Chinese population | July 1, 2020 to December 31, 2025
  Clearance (CL) will be calculated through multiple plasma concentrations drawn from the patients after taking venetoclax.

SECONDARY OUTCOMES:
Analysis of venetoclax plasma concentration with concomitant CYP enzyme inhibitors or inducers | July 1, 2020 to December 31, 2025
  Concomitant CYP enzyme inhibitors or inducers of each patients will be recorded and analyzed its actual impact on venetoclax pharmacokinetic parameters.
Association between venetoclax plasma concentration and therapeutic effectiveness, adverse events | July 1, 2020 to December 31, 2025
  The relationship between venetoclax plasma concentration and its therapeutic effectiveness, adverse events will be investigated during continuous follow-ups this study.
Establishment of venetoclax clinical dose adjustment | July 1, 2020 to December 31, 2025
  Identify the concentration cut-off points of effectiveness and toxicity respectively, and validate these cut-off points externally in future clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No